CLINICAL TRIAL: NCT06398782
Title: The Impact of DXA-Based Body Composition Phenotypes on the All-cause Mortality Among the US Cancer Survivors
Brief Title: Prognostic Effect of Body Composition in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Director, West China Hospital
Other Study IDs: #98-12, #2005-06, #2011-17
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Body Composition; Morality; Cancer Survivor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 230 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: body composition assessment — body composition of cancer survivors were assessed by Dual-energy X-ray absorptiometry

SUMMARY:
This study aims to evaluate the association between body composition and mortality risk among the US population based on data from the National Health and Nutrition Examination Survey (NHANES), a nationally representative cohort.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cancer diagnosis beyond 18 years old.

Exclusion Criteria:

* Participants with missing cancer investigations and incomplete DXA body composition data were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data were extracted from National Health and Nutrition Examination Survey (NHANES) 1999 to 2006 and 2011 to 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality | Jan 1 1999 to Dec 31 2019
  To evaluate the association between fat mass index (FMI, fat mass and height will be combined to report FMI in kg/m^2) and all-cause mortality among cancer survivors.
Rate of all-cause mortality | Jan 1 1999 to Dec 31 2019
  To evaluate the association between muscle mass index (MMI, muscle mass and height will be combined to report MMI in kg/m^2) and all-cause mortality among cancer survivors.